CLINICAL TRIAL: NCT02017964
Title: A Phase II Study for the Treatment of Non-metastatic Nodular Desmoplastic Medulloblastoma in Children Less Than 4 Years of Age
Brief Title: Combination Chemotherapy in Treating Younger Patients With Newly Diagnosed, Non-metastatic Desmoplastic Medulloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS1221; NCI-2013-02379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ACNS1221; ACNS1221; s15-00476; ACNS1221 (Other: Children's Oncology Group); ACNS1221 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2013-12-13; First posted 2013-12-23 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Desmoplastic/Nodular Medulloblastoma; Medulloblastoma; Medulloblastoma With Extensive Nodularity; Nevoid Basal Cell Carcinoma Syndrome
MeSH Terms: conditions — Medulloblastoma; Basal Cell Nevus Syndrome | interventions — Carboplatin; Mental Status and Dementia Tests; Cyclophosphamide; Etoposide; Methotrexate; merphos; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): INDUCTION THERAPY: Patients receive vincristine sulfate IV over 1 minute or infused via minibag on days 1, 15, and 29; cyclophosphamide IV over 1 hour on days 1-3; methotrexate IV over 24 hours on days 15 and 29; etoposide IV over 60-120 minutes on days 43-45; and carboplatin IV over 1 hour on days 43-45. Treatment repeats every 63 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  CONTINUATION THERAPY: Patients receive vincristine sulfate IV over 1 minute or infused via minibag on day 1, cyclophosphamide IV over 1 hour on days 1-3, etoposide IV over 60-120 minutes on days 21-23, and carboplatin IV over 1 hour on days 21-23. Treatment repeats every 42 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Cognitive Assessment; Drug: Cyclophosphamide; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Cognitive Assessment — Optional ancillary studies
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well combination chemotherapy works in treating younger patients with newly diagnosed, non-metastatic desmoplastic medulloblastoma. Drugs used in chemotherapy, such as vincristine sulfate, cyclophosphamide, methotrexate, etoposide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate of the progression free survival (PFS) distribution for patients 0-<4 years of age with M0 desmoplastic medulloblastoma (nodular desmoplastic or medulloblastoma with extensive nodularity) treated with the modified HIT SKK regimen (excluding the use of intraventricular methotrexate).

OTHER PRE-SPECIFIED OBJECTIVES:

I. Evaluate the feasibility of a rapid central pathology screening review for treatment allocation according to histology and assess agreement between institutional and central pathology review diagnoses as well as among central pathology review diagnoses.

II. Prospectively evaluate the molecular profile of nodular desmoplastic (ND)/medulloblastoma with extensive nodularity (MBEN) medulloblastoma in young children.

III. Monitor and describe the neurocognitive and adaptive functioning of young children with ND/MBEN medulloblastoma treated on this protocol using the ALTE07C1 protocol.

OUTLINE:

INDUCTION THERAPY: Patients receive vincristine sulfate intravenously (IV) over 1 minute or infused via minibag on days 1, 15, and 29; cyclophosphamide IV over 1 hour on days 1-3; methotrexate IV over 24 hours on days 15 and 29; etoposide IV over 60-120 minutes on days 43-45; and carboplatin IV over 1 hour on days 43-45. Treatment repeats every 63 days for 3 courses in the absence of disease progression or unacceptable toxicity.

CONTINUATION THERAPY: Patients receive vincristine sulfate IV over 1 minute or infused via minibag on day 1, cyclophosphamide IV over 1 hour on days 1-3, etoposide IV over 60-120 minutes on days 21-23, and carboplatin IV over 1 hour on days 21-23. Treatment repeats every 42 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 16, 20, 24, 36, 48, 60, and 72 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed and have a confirmed histologic diagnosis of nodular desmoplastic (ND) medulloblastoma or medulloblastoma with extensive nodularity (MBEN) from rapid central pathology screening review; please note: patients with Gorlin syndrome are eligible
* Patient must have negative lumbar cerebrospinal fluid (CSF) cytology (lumbar CSF must be obtained unless medically contraindicated); CSF cytology for staging should be performed preferably no sooner than 14 days post operatively to avoid false positive CSF, ideally, CSF should be obtained between day 14 and day 21 to allow for final staging status before enrollment onto the study; Note: patients with positive CSF cytology obtained prior to 14 days after surgery may have cytology repeated to determine eligibility and final CSF status
* Patients must have:

  * Pre-operative cranial magnetic resonance imaging (MRI) (recommended with gadolinium) or pre-operative computed tomography (CT) (recommended with contrast)
  * Post-operative cranial MRI with and without gadolinium within 72 hours of surgery
  * Spinal MRI pre-op with and without gadolinium or post-op with and without gadolinium preferably within 72 hours of surgery
* Patients must be enrolled on study within 31 days of definitive surgical resection at which time tissue is acquired to determine a diagnosis; patients must be enrolled before treatment begins; the date protocol therapy is projected to start must be no later than five (5) calendar days after the date of study enrollment; patients who are started on protocol therapy on a Phase II study prior to study enrollment will be considered ineligible
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Patients who are receiving dexamethasone must be on a stable dose for at least 1 week prior to study entry
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 10.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age
* Central nervous system function defined as:

  * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
  * Patients must not be in status, coma or assisted ventilation prior to study enrollment

Exclusion Criteria:

* Patients with metastatic disease by either MRI evaluation (brain and spine) or lumbar CSF cytology are not eligible
* Patients must not have received any prior tumor-directed therapy other than surgical intervention and corticosteroids

Max Age: 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2013-12-24 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie E Lafay-Cousin, Principal Investigator — Children's Oncology Group
Locations (173):
- United States (158):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened for entry on December 24, 2013, and the first patient was enrolled on April 22, 2014. The study enrolled 26 patients before being closed early due to inferior efficacy as of July 27, 2016. 25 of the 26 patients enrolled were deemed to be eligible
Groups:
- All Patients (Combination Chemotherapy): All patients enrolled on the study. Patients received 3-5 cycles of therapy which included cyclophosphamide (800 mg/m2/day), vincristine (1.5 mg/m2/day), methotrexate (5,000 mg/m2), etoposide (150 mg/m2/dose) and carboplatin (200 mg/m2/day IV).
Period: Overall Study
Arm/Group | All Patients (Combination Chemotherapy)
Started | 26
Completed | 25
Not Completed | 1
Not completed — Patient deemed ineligible | 1

BASELINE CHARACTERISTICS:
Groups:
- All Eligible Patients (Combination Chemotherapy): All eligible patients enrolled on the study
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: months (at time of dx)] | 19.7 [7.1 to 42.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 23
  Canada | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time interval from diagnosis to the earliest of disease progression/recurrence or death from any cause, or to the date of last follow-up for patients without events. PFS was estimated using the method of Kaplan and Meier. 2-year estimates are reported with 95% CI's.
Time Frame: 2 years from diagnosis
Population: 26 patients were enrolled on the protocol, but 1 was deemed ineligible. The ineligible patient was excluded from all analyses.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 25
percent probability | 52.0 [32.4 to 71.6]

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from diagnosis to death from any cause, or to the date of last follow-up for survivors. OS was estimated using the method of Kaplan and Meier. 2-year estimates are reported with 95% CI's, as the data are not mature to 72 months.
Time Frame: Assessed up to 72 months, reported at 2 years from diagnosis
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 25
percent probability | 92.0 [80.8 to 100.0]

3. Primary Outcome: Event-free Survival (EFS)
Description: Event-free survival (EFS) is defined as the time from diagnosis to the earliest of disease progression/recurrence, second malignancy or death from any cause, or to the date of last follow-up for patients without events. EFS was estimated using the method of Kaplan and Meier. 2-year estimates are reported with 95% CI's.
Time Frame: 2 years from diagnosis
Population: 26 patients were enrolled on the protocol, but 1 was deemed ineligible. The ineligible patient is excluded from all analyses.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 25
percent probability | 52.0 [32.4 to 71.6]

4. Primary Outcome: Percentage of Patients With Responses at 189 Days
Description: The percentage of patients with complete response (CR) at the end of induction (~189 days) was reported and presented with the associated exact 95% confidence interval.
Time Frame: 189 days from start of treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 25
Percentage of patients | 92.0 [75.6 to 98.6]

5. Primary Outcome: Percentage of Patients With Responses at 273 Days
Description: The percentage of patients with complete response (CR) at the end of therapy (~273 days) was reported and presented with the associated exact 95% confidence interval.
Time Frame: 273 days from start of treatment
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | All Eligible Patients (Combination Chemotherapy)
Number analyzed (Participants) | 25
Percentage of patients | 88.0 [69.7 to 96.7]

6. Other Pre Specified Outcome: Feasibility of Rapid Central Pathology Screening Review Defined as Success Rate of Timely Central Pathology Review Based on the Expectation That at Least 95% of the Cases Will be Reviewed Within 10 Days
Description: At the end of the trial the feasibility of such a prescreening process will be assessed by reporting the percentage and the associated confidence interval of cases where the central review was obtained within 10 days from receipt of slides.
Time Frame: Up to 10 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Molecular Profile
Description: Contingency table analysis will be used to examine the association of molecular profile with histology.
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Neurocognitive and Adaptive Functioning Assessed Using Full Scale IQ Score (FSIQ) and General Adaptive Composite Score (GAC)
Description: Changes will be described via paired tests and confidence intervals both for FSIQ and GAC in order to capture any deterioration over time.
Time Frame: Baseline to up to 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event reporting is collected routinely using case report forms. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | All Eligible Patients (Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Eligible Patients (Combination Chemotherapy) (N=25)
Death NOS (General disorders) | 1 (1)
Other, Progression Of Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Eligible Patients (Combination Chemotherapy) (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (4)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (18)
Neutrophil count decreased (Investigations) | 14 (36)
Platelet count decreased (Investigations) | 7 (13)
White blood cell decreased (Investigations) | 11 (24)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT02017964/Prot_SAP_000.pdf